CLINICAL TRIAL: NCT07188454
Title: Intervention Programs and Outcomes for Managing Behavioral Problems in Dementia
Brief Title: The Effects of a Meditation Intervention on the Psychological Burden of Long-Term Care Professionals and Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC1110102-R4
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Burnout, Professional; Caregivers; Caregivers Burnout; Stress, Psychological
Keywords: Meditation; Mindfulness; Digital health intervention; Caregiver burnout; Caregiver burden; Professional caregivers; Family caregivers; Stress reduction; Mental health; Randomized controlled trial
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Caregiver Burden; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Meditation Intervention (Experimental): Participants received a 5-week digitally supported mindfulness program immediately after randomization. The program included five weekly 90-minute live online classes led by an instructor and daily guided mindfulness practice (about 10 minutes per day) using the AIZEN digital platform, with automated reminders delivered via the LINE messaging service.
  Interventions: Behavioral: Mindfulness-Based Digital Intervention (AIZEN Program)
- Wait-list Control (No Intervention): Participants were assigned to a wait-list control condition and did not receive the intervention during the first 5 weeks after randomization. After completing post-intervention assessments at Week 5, they received the identical 5-week mindfulness program, consisting of weekly 90-minute live online classes and daily guided mindfulness practice with the AIZEN platform.

INTERVENTIONS:
Behavioral: Mindfulness-Based Digital Intervention (AIZEN Program) — The intervention consisted of a 5-week mindfulness program designed for caregivers. Participants attended one live, instructor-led online class each week (90 minutes per session) delivered via Microsoft Teams. Between classes, they were asked to complete at least 10 minutes of daily guided mindfulness practice using the AIZEN digital platform. To encourage adherence, participants also received automated daily reminders through the LINE messaging service.
  Arms: Immediate Meditation Intervention

SUMMARY:
The goal of this clinical trial is to learn whether a brief, digitally-supported mindfulness program can reduce caregiver burnout in professional caregivers (such as nurses, case managers, and care workers) and informal family caregivers in Taiwan.

The main questions it aims to answer are:

Does the mindfulness program reduce personal and work-related burnout among professional caregivers?

Does the mindfulness program reduce caregiver burden among informal family caregivers?

Researchers compared an immediate-intervention group with a wait-list control group to see if those who received the program earlier experienced greater improvements.

Participants were asked to:

Join five weekly 90-minute live online classes led by an instructor.

Practice daily 10-minute guided mindfulness sessions using the AIZEN digital platform.

Complete questionnaires about stress and caregiver burden at three time points: baseline (T1), after the 5-week program (T2), and 5-week follow-up (T3).

DETAILED DESCRIPTION:
This study was a randomized, stratified, wait-list-controlled pilot clinical trial conducted in Taiwan to evaluate the feasibility and preliminary efficacy of a digitally-supported mindfulness program for caregivers.

Participants were randomized 1:1 to either:

Immediate-intervention group (received the 5-week program immediately after randomization), or

Wait-list control group (received the same program after completing their post-intervention assessment at 5 weeks).

Participants were stratified by caregiver type (professional vs. informal), age (younger vs. older than the sample median), and perceived stress level (low vs. high). Randomization was computer-generated and implemented independently of outcome assessment.

The intervention was a 5-week program consisting of:

Weekly 90-minute live, instructor-led sessions delivered via Microsoft Teams.

Daily home practice supported by guided meditation audio tracks on the AIZEN digital platform.

Automated daily reminders through the LINE messaging service to encourage adherence.

Outcome assessments were collected at three time points:

T1 (Baseline, Week 0) - prior to randomization

T2 (Post-intervention, Week 5) - after completion of the immediate group's program

T3 (Follow-up, Week 10) - after the wait-list group completed the program

The primary outcomes were changes in burnout among professional caregivers, assessed with the Chinese version of the Copenhagen Burnout Inventory (CBI), including personal, work-related, and client-related dimensions. A secondary exploratory outcome was caregiver burden among informal caregivers, assessed with the Zarit Burden Interview (ZBI).

Statistical analyses used linear mixed-effects models with planned contrasts to evaluate three core hypotheses:

Primary intervention effect: whether changes from T1 to T2 differed between groups (difference-in-differences).

Replication effect: whether the wait-list group showed improvements after receiving the program (T2 to T3).

Maintenance effect: whether benefits for the immediate-intervention group were sustained at follow-up (T2 to T3).

In addition, exploratory analyses included adjustment for work over-commitment as a covariate and evaluation of whether daily home practice (logged via the AIZEN platform) mediated intervention effects.

This study was designed as a feasibility and proof-of-concept trial to inform the scalability of digital mindfulness interventions for caregivers in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Currently engaged in paid professional caregiving (e.g., nurse, care worker, case manager) or unpaid informal/family caregiving
* Able to attend weekly online sessions via Microsoft Teams
* Willing to complete web-based questionnaires
* Willing to undertake at least 10 minutes of daily mindfulness practice
* No prior meditation experience within the three months preceding recruitment

Exclusion Criteria:

* Did not meet the definition of caregiver (professional or informal)
* Prior meditation practice within the three months before recruitment
* Unwilling or unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-09-13 (Actual)

PRIMARY OUTCOMES:
Change in Personal Burnout (Copenhagen Burnout Inventory, Professional Caregivers) | Baseline (Week 0), Post-intervention (Week 5), and Follow-up (Week 10)
  Personal burnout was measured using the Chinese version of the Copenhagen Burnout Inventory (CBI). This subscale includes 5 items that assess general physical and psychological exhaustion. Each item is scored on a 5-point scale (0 = "never" to 100 = "always"), and the subscale score is calculated as the mean of all items, with higher scores indicating greater burnout.
Change in Work-Related Burnout (Copenhagen Burnout Inventory, Professional Caregivers) | Baseline (Week 0), Post-intervention (Week 5), and Follow-up (Week 10)
  Work-related burnout was measured using the Chinese version of the Copenhagen Burnout Inventory (CBI). This subscale consists of 5 items that assess exhaustion specifically attributed to work demands. Each item is scored on a 5-point scale (0 = "never" to 100 = "always"), and the subscale score is calculated as the mean of all items, with higher scores indicating greater burnout.
Change in Client-Related Burnout (Copenhagen Burnout Inventory, Professional Caregivers) | Baseline (Week 0), Post-intervention (Week 5), and Follow-up (Week 10)
  Client-related burnout was measured using the Chinese version of the Copenhagen Burnout Inventory (CBI). This subscale consists of 6 items that assess exhaustion specifically attributed to interactions with care recipients or clients. Each item is scored on a 5-point scale (0 = "never" to 100 = "always"), and the subscale score is calculated as the mean of all items, with higher scores indicating greater burnout.

SECONDARY OUTCOMES:
Change in Caregiver Burden (Zarit Burden Interview, Informal Caregivers) | Baseline (Week 0), Post-intervention (Week 5), and Follow-up (Week 10)
  Caregiver burden was measured using the Chinese version of the Zarit Burden Interview (ZBI). This validated instrument consists of 22 items that assess the impact of caregiving on the caregiver's emotional, social, and physical well-being. Each item is rated on a 5-point scale (0 = "never" to 4 = "nearly always"), with total scores ranging from 0 to 88. Higher scores indicate greater caregiver burden.

CONTACTS AND LOCATIONS:
Locations (1):
- National Health Research Institutes, Zhunan, Taiwan

IPD SHARING:
Plan to Share IPD: No